CLINICAL TRIAL: NCT00820170
Title: A Phase I-II Study of Dasatinib in Combination With Weekly Paclitaxel for Patients With Metastatic Breast Carcinoma
Brief Title: Dasatinib In Combination With Weekly Paclitaxel For Patients With Metastatic Breast Carcinoma CA 180 194
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-122
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: Breast; Cancer; DASATINIB; TAXOL (PACLITAXEL); 08-122
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Dasatinib; Paclitaxel

ARMS (1):
- dasatinib and paclitaxel (Experimental): The phase I portion is a standard, three-patient per cohort, dose escalation schedule will be used. Between 6 and 54 patients will likely be necessary to determine the MTD of dasatinib in combination with weekly paclitaxel.
  The phase II portion of this trial has a Simon two-stage design to determine the efficacy of dasatinib when administered in combination with paclitaxel.
  Interventions: Drug: Dasatinib and Paclitaxel

INTERVENTIONS:
Drug: Dasatinib and Paclitaxel — A treatment cycle will consist of 28 days, according to the following schedule:
  Dasatinib 120MG PO once daily, Weekly paclitaxel 80 mg/m2 given intravenously over 1 hour on day 1, 8, and 15 of a 28 day cycle.
  The trial will initially test the combination of weekly paclitaxel and dasatinib given PO, once daily , continuously. In case of 2 dose-limiting toxicities (DLT) in the first cohort (0), the next cohort will test dasatinib given with a different schedule, 5 days on and 2 days off, omitting dasatinib the day prior and the day of administration of paclitaxel.

SUMMARY:
The purpose of this study is to find the highest dose of dasatinib that can be safely given to a patient when the drug is given in combination with the known anticancer drug paclitaxel. Paclitaxel is an established anti-cancer drug, used in the treatment of many cancers, and it is an approved treatment for breast cancer. Dasatinib has been approved by the Food and Drug Administration for use as a single therapy in another kind of cancer, but its use in breast cancer patients, and in combination with paclitaxel is investigational.

In this study, we will test the safety of dasatinib when given at different dose levels in combination with paclitaxel. We want to find out what effects, good and/or bad, it has on the patient and on metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients with diagnosis of invasive adenocarcinoma of the breast confirmed at MSKCC.
* For the phase I portion, patients with any ER/PR/HER2 disease status, no longer eligible for hormonal therapy or HER2-targeted therapy, will be eligible.
* For the phase II portion, there needs to be documentation of negative HER2 (IHC 0-1+ or FISH/CISH negative) status. Patients with any ER/PR disease status are eligible.
* A paraffin-embedded tissue block or unstained slides from prior surgery must be available.
* Evidence of recurrent or progressive locally advanced or metastatic breast cancer.

Presence of:

* For the phase I portion: at least one evaluable or measurable metastatic lesion ,
* For the phase II portion: at least one measurable metastatic lesion according to the RECIST criteria which has not been irradiated (i.e. newly arising lesions in previously irradiated areas are accepted). Ascites, pleural effusion, and bone metastases are not considered measurable. Minimum indicator lesion size: > or = to 10 mm measured by spiral CT or > or = to 20 mm measured by conventional techniques.

Prior therapies:

For the phase I portion: Any number of prior endocrine or biologic therapies is permitted . In addition, patients may be untreated in the metastatic setting or have received any number of prior cytotoxic regimens.

For the phase II portion: 0-2 prior therapies for metastatic disease are allowed.

Prior taxane therapy, either in the adjuvant or in the metastatic setting, either deliver weekly, q 2 weeks or q 3 weeks, will be permitted. Prior therapy with bevacizumab will be allowed. All previous chemotherapy, radiotherapy and intravenous biphosphonates must have been discontinued at least 3 weeks prior to study entry, 3 weeks also for trastuzumab and bevacizumab. All acute toxic effects (excluding alopecia) of any prior therapy must have resolved to NCI CTC (Version 3) Grade ≤1.

* Endocrine therapy with an aromatase inhibitor, SERM (ie, tamoxifen) or fulvestrant is permitted, however it must be discontinued before enrolling in the study.
* ECOG performance status of 0 or 1.
* Age > or = to 18 years old. Adequate Organ Function
* Total bilirubin ≤ 1.5 times the institutional Upper Limit of Normal (ULN)
* Hepatic enzymes (AST, ALT ) ≤ 2.5 times the institutional ULN
* Serum Na, K+, Mg2+, Phosphate and Ca2+≥ Lower Limit of Normal (LLN)
* Serum Creatinine ≤ 1.5 time the institutional ULN
* Neutrophil count, Platelets, both Grade 0-1
* PT (INR) and PTT Grade 0-1, except for patients on Coumadin or low molecular weight heparin
* Ability to take oral medication (dasatinib must be swallowed whole)

Concomitant Medications:

* Patient agrees to discontinue St. Johns Wort while receiving dasatinib therapy
* Patient agrees that IV biphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia. Concomitant Medications, any of the following should be considered for exclusion:

Patient agrees to discontinue QT-prolonging agents strongly associated with Torsades de Pointes including: (patients must discontinue drug ≥ 7 days prior to starting dasatinib) such as:

* quinidine, procainamide, disopyramide
* amiodarone, sotalol, ibutilide, dofetilide
* erythromycin, clarithromycin
* chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
* cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.
* The concomitant use of H2 blockers or proton pump inhibitors with dasatinib is not recommended. The use of antacids should be considered in place of H2 blockers or proton pump inhibitors in patients receiving dasatinib therapy. If antacid therapy is needed, the antacid dose should be administered at least 2 hours prior to or 2 hours after the dose of dasatinib.
* Patient may not be receiving any potent CYP3A4 inhibitors. These are prohibited (patients must discontinue drug ≥7 days prior to starting dasatinib) and include:
* itraconazole, ketoconazole, miconazole, coriconazole
* amprenavir, atazanavir, fosamprenavir, indinavir, nelfinavir, ritonavir
* ciprofloxacin, clarithromycin, diclofenac, doxycycline, enoxacin, imatinib, isoniazid
* ketamine, nefazodone, nicardipine, propofol, quinidine, telithromycin

Women of childbearing potential (WOCBP) must have:

* A negative serum or urine pregnancy test within 72 hours prior to the start of study drug administration
* Persons of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 4 weeks after study drug is stopped
* Pregnant or nursing women may not participate. Patients of reproductive potential may not participate unless they have agreed to use an effective method of contraception and to continue contraception for 30 days from the date of the last study drug administration. Postmenopausal woman must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Signed written informed consent including a HIPAA form according to institutional guidelines.

Exclusion Criteria:

* Life expectancy < 3 months.
* Prior severe allergic reaction to paclitaxel therapy.
* Presence of new or recurrent pleural effusion which is symptomatic and/or requiring medical intervention (NCI CTC Grade 2, 3 or 4).
* Completion of previous chemotherapy regimen < 3 weeks prior to the start of study treatment.
* Prior hormonal therapy must be discontinued prior to treatment start. Biologic therapy (eg, bevacizumab, trastuzumab) for the treatment of metastatic disease must be discontinued > or = to 3 weeks from the start of protocol treatment.

Concurrent medical condition which may increase the risk of toxicity.

Patients may not have any clinically significant cardiovascular disease including the following:

* myocardial infarction or ventricular tachyarrhythmia within 6 months
* prolonged QTc >480 msec (Fridericia correction)
* ejection fraction less than institutional normal
* major conduction abnormality (unless a cardiac pacemaker is present)
* Patients with any cardiopulmonary symptoms of unknown cause (e.g. shortness of breath, chest pain, etc.) should be evaluated by a baseline echocardiogram with or without stress test as needed in addition to electrocardiogram (EKG) to rule out QTc prolongation. The patient may be referred to a cardiologist at the discretion of the principal investigator. Patients with underlying cardiopulmonary dysfunction should be excluded from the study.
* Subjects with hypokalemia or hypomagnesemia if it cannot be corrected prior to dasatinib administration

History of significant bleeding disorder unrelated to cancer, including:

Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)

* Diagnosed acquired bleeding disorder within one year (e.g., acquired antifactor VIII antibodies)
* Ongoing or recent (≤ 3 months) significant gastrointestinal bleeding Other medical condition which in the opinion of the Investigator might confer an unacceptable increase in risk.
* Patients with symptomatic CNS metastases that remain untreated by radiation therapy are excluded from this trial. The presence of asymptomatic brain metastases or brain metastases that have been previously irradiated are not grounds for trial exclusion.
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake.
* Presence of uncontrolled gastrointestinal malabsorption syndrome.
* Unwillingness to give written informed consent or unwillingness to participate or inability to comply with the protocol for the duration of the study. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures are necessary for participation in this clinical trial.
* Concurrent radiotherapy is not permitted for disease progression on treatment on protocol, but might allowed for pre-existing non-target lesions with approval from the principal investigator of the trial.
* Patients with > Grade 1 neuropathy will be excluded form this trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-01; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Fornier, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 100 mg: Paclitaxel 80 mg/m2 weekly 3/4; Dasatinib 100 mg daily continuously
- Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 150 mg: Paclitaxel 80 mg/m2 weekly 3/4; Dasatinib 150 mg daily continuously
- Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 70 mg: Paclitaxel 80 mg/m2 weekly 3/4; Dasatinib 70 mg daily continuously
- Phase 2: Paclitaxel 80 mg/m2 + Dasatinib 120 mg: Paclitaxel 80 mg/m2 weekly 3/4; Dasatinib 120 mg daily continuously
- Participants Who Did Not Receive Treatment: Participants did not receive treatment
Period: Overall Study
Arm/Group | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 100 mg | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 150 mg | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 70 mg | Phase 2: Paclitaxel 80 mg/m2 + Dasatinib 120 mg | Participants Who Did Not Receive Treatment
Started | 3 | 5 | 3 | 40 | 4
Completed | 3 | 5 | 3 | 40 | 0
Not Completed | 0 | 0 | 0 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The 3 participants treated in the Phase I portion of the study at Paclitaxel 80mg/m2 + Dasatinib 120 mg were included in the group of 40 participants in the Phase II portion of this study.
Groups:
- No Arm Selected: No Treatment Arm Selected
- Total: Total of all reporting groups
Arm/Group | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 100 mg | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 150 mg | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 70 mg | Phase 2: Paclitaxel 80 mg/m2 + Dasatinib 120 mg | No Arm Selected | Total
Number analyzed (Participants) | 3 | 5 | 3 | 40 | 4 | 55
Age, Continuous [Mean (Full Range); unit: years] | 53 [39 to 67] | 56 [41 to 74] | 59 [54 to 62] | 50.7 [30 to 79] | 52.5 [47 to 58] | 51.89 [30 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 3 | 37 | 4 | 52
  Male | 0 | 0 | 0 | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 5 | 0 | 7
  White | 3 | 4 | 2 | 32 | 2 | 43
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 5 | 3 | 40 | 4 | 55

OUTCOME MEASURES:

1. Primary Outcome: Phase I Portion: Maximum Tolerated Dose/MTD of Dasatinib When Administered in Combination With a Fixed Dose of Weekly Paclitaxel.
Time Frame: Through completion of Phase I, up to 1 year
Population: 15 participants were enrolled for the Phase I portion of the study. These 15 participants determined the MTD for the study.
Measure: Number; unit: mg of dasatinib
Groups:
- Dasatinib and Paclitaxel: The phase I portion is a standard, three-patient per cohort, dose escalation schedule will be used. Between 6 and 54 patients will likely be necessary to determine the MTD of dasatinib in combination with weekly paclitaxel.
  The phase II portion of this trial has a Simon two-stage design to determine the efficacy of dasatinib when administered in combination with paclitaxel.
  Dasatinib and Paclitaxel: A treatment cycle will consist of 28 days, according to the following schedule:
  Dasatinib 120MG PO once daily, Weekly paclitaxel 80 mg/m2 given intravenously over 1 hour on day 1, 8, and 15 of a 28 day cycle.
  The trial will initially test the combination of weekly paclitaxel and dasatinib given PO, once daily , continuously. In case of 2 dose-limiting toxicities (DLT) in the first cohort (0), the next cohort will test dasatinib given with a different schedule, 5 days on and 2 days off, omitting dasatinib the day prior and the day of administration of paclitaxel.
Arm/Group | Dasatinib and Paclitaxel
Number analyzed (Participants) | 15
mg of dasatinib | 120

2. Primary Outcome: Efficacy (Objective Response Rate; ORR; Complete Response (CR) + Partial Response (PR)) of Dasatinib When Administered in Combination With Weekly Paclitaxel at the MTD Established During the Phase I Portion of This Trial.
Time Frame: Through study completion, up to 2 years
Population: The 3 participants treated in the Phase I portion of the study at Paclitaxel 80mg/m2 + Dasatinib 120 mg were included in the group of 40 participants in the Phase II portion of this study. Results and data analysis reflect this.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 100 mg | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 150 mg | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 70 mg | Phase 2: Paclitaxel 80 mg/m2 + Dasatinib 120 mg | No Arm Selected
Number analyzed (Participants) | 3 | 5 | 3 | 40 | 4
Participants
  Stable Disease | 3 | 1 | 1 | 15 | 1
  Complete Response | 0 | 0 | 0 | 1 | 0
  Partial Response | 0 | 1 | 0 | 10 | 0
  Progression of Disease | 0 | 2 | 2 | 10 | 1
  Not Evaluable for Response | 0 | 1 | 0 | 4 | 2

3. Secondary Outcome: Median Overall Survival for Phase II Participants
Description: Overall Survival for Phase II Participants
Time Frame: Through study completion, up to 2 years
Population: This objective is specific for the Phase II participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 100 mg | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 150 mg | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 70 mg | Phase 2: Paclitaxel 80 mg/m2 + Dasatinib 120 mg | No Arm Selected
Number analyzed (Participants) | 0 | 0 | 0 | 40 | 0
months |  |  |  | 20.6 [12.9 to 25.2] |

4. Secondary Outcome: Participant Adverse Events to Measure Safety and Tolerability of Dasatinib When Administered in Combination With Weekly Paclitaxel.
Description: Evaluate adverse events using CTCAE v3
Time Frame: Through study completion, up to 2 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: Paclitaxel 80 mg/m2 + Dasatinib 100 mg: Paclitaxel 80 mg/m2 weekly 3/4; Dasatinib 100 mg daily continuously
- Arm 2: Paclitaxel 80 mg/m2 + Dasatinib 120 mg: Paclitaxel 80 mg/m2 weekly 3/4; Dasatinib 120 mg daily continuously
- Arm 3: Paclitaxel 80 mg/m2 + Dasatinib 150 mg: Paclitaxel 80 mg/m2 weekly 3/4; Dasatinib 150 mg daily continuously
- Paclitaxel 80 mg/m2 + Dasatinib 70 mg: Paclitaxel 80 mg/m2 weekly 3/4; Dasatinib 70 mg daily continuously
Arm/Group | Arm 1: Paclitaxel 80 mg/m2 + Dasatinib 100 mg | Arm 2: Paclitaxel 80 mg/m2 + Dasatinib 120 mg | Arm 3: Paclitaxel 80 mg/m2 + Dasatinib 150 mg | Paclitaxel 80 mg/m2 + Dasatinib 70 mg | No Arm Selected
Number analyzed (Participants) | 3 | 40 | 5 | 3 | 4
Participants | 3 | 40 | 5 | 3 | 4

5. Secondary Outcome: Median Progression Free Survival for Phase II Participants
Description: Per RECIST criteria, Progression (PD) is defined at least a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Through study completion, up to 2 years
Population: This objective is specific for the Phase II participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 100 mg | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 150 mg | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 70 mg | Phase 2: Paclitaxel 80 mg/m2 + Dasatinib 120 mg | No Arm Selected
Number analyzed (Participants) | 0 | 0 | 0 | 40 | 0
months |  |  |  | 5.2 [2.9 to 9.9] |

6. Secondary Outcome: Phase II: Number of Participants With Clinical Benefit According to Tumor Biomarker Data: Assays of VEGFR2
Description: Tumor biomarker data obtained at baseline and after 2 cycles of treatment (8 weeks), will be performed by enzyme-linked immunosorbent assay. Clinical Benefit is defined as the sum of the percentage of participants who achieved CR, PR and stable disease for > 6 months.
Time Frame: 8 weeks
Population: Phase II participants only
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 100 mg | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 150 mg | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 70 mg | Phase 2: Paclitaxel 80 mg/m2 + Dasatinib 120 mg | No Arm Selected
Number analyzed (Participants) | 0 | 0 | 0 | 40 | 0
Participants
  Discontinued prior to 1st Assessment | 0 | 0 | 0 | 5 | 0
  Clinical Benefit, VEGF collected | 0 | 0 | 0 | 13 | 0
  No Clinical Benefit, VEGF Collected | 0 | 0 | 0 | 19 | 0
  Clinical Benefit, VEGF Not Collected | 0 | 0 | 0 | 2 | 0
  No Clinical Benefit, VEGF Not Collected | 0 | 0 | 0 | 1 | 0

7. Secondary Outcome: Median Time To Progression for Phase II Participants
Time Frame: Through study completion, up to 2 years
Population: This objective is specific for the Phase II participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 100 mg | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 150 mg | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 70 mg | Phase 2: Paclitaxel 80 mg/m2 + Dasatinib 120 mg | No Arm Selected
Number analyzed (Participants) | 0 | 0 | 0 | 40 | 0
months |  |  |  | 5.84 [0 to 25.7] |

8. Secondary Outcome: Phase II: Number of Participants With Clinical Benefit According to Circulating Tumor Cells (CTC) at Baseline and After 2 Cycles of Treatment (8 Weeks)
Description: Phase II participants only
Time Frame: 8 weeks
Population: Phase II participants only
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 100 mg | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 150 mg | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 70 mg | Phase 2: Paclitaxel 80 mg/m2 + Dasatinib 120 mg | No Arm Selected
Number analyzed (Participants) | 0 | 0 | 0 | 40 | 0
Participants
  Discontinued treatment prior to 1st assessment | 0 | 0 | 0 | 5 | 0
  Clinical Benefit, CTC Collection | 0 | 0 | 0 | 14 | 0
  No Clinical Benefit, CTC Collection | 0 | 0 | 0 | 20 | 0
  Clinical Benefit, No CTC Collected | 0 | 0 | 0 | 1 | 0

9. Secondary Outcome: Phase II: Exploratory Somatic Gene Mutations Detection in Archived Tumor Samples
Time Frame: 2 years
Population: Data were not collected
Arm/Group | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 100 mg | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 150 mg | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 70 mg | Phase 2: Paclitaxel 80 mg/m2 + Dasatinib 120 mg | No Arm Selected
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Phase I: 1 year Phase II: 2 years
Description: 3 participants treated in the Phase I portion of the study at Paclitaxel 80mg/m2 + Dasatinib 120 mg were included in the group of 40 participants in the Phase II portion of this study.
Groups:
- Phast 1: Paclitaxel 80 mg/m2 + Dasatinib 70 mg: Paclitaxel 80 mg/m2 weekly 3/4; Dasatinib 70 mg daily continuously
Arm/Group | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 100 mg | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 150 mg | Phast 1: Paclitaxel 80 mg/m2 + Dasatinib 70 mg | Phase 2: Paclitaxel 80 mg/m2 + Dasatinib 120 mg | No Arm Selected
All-Cause Mortality (participants affected / at risk) | 3/3 | 5/5 | 3/3 | 5/40 | 4/4
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/5 | 0/3 | 11/40 | 0/4
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 2/3 | 40/40 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 100 mg (N=3) | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 150 mg (N=5) | Phast 1: Paclitaxel 80 mg/m2 + Dasatinib 70 mg (N=3) | Phase 2: Paclitaxel 80 mg/m2 + Dasatinib 120 mg (N=40) | No Arm Selected (N=4)
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0
Hemoglobin decreased/Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Laboratory test abnormal (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 100 mg (N=3) | Phase 1: Paclitaxel 80 mg/m2 + Dasatinib 150 mg (N=5) | Phast 1: Paclitaxel 80 mg/m2 + Dasatinib 70 mg (N=3) | Phase 2: Paclitaxel 80 mg/m2 + Dasatinib 120 mg (N=40) | No Arm Selected (N=4)
ALT, SGPT (Investigations) | 1 | 1 | 0 | 6 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0
Hyperbilirubinemia (Investigations) | 1 | 1 | 0 | 2 | 0
Creatinine (Investigations) | 1 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0 | 8 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 7 | 0
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 11 | 0
Heartburn/Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Hemoglobin (Blood and lymphatic system disorders) | 1 | 3 | 0 | 19 | 0
INR (Investigations) | 1 | 0 | 1 | 1 | 0
Infection, other (Infections and infestations) | 1 | 1 | 0 | 0 | 0
White Blood Cells/Leukocytes (Investigations) | 1 | 3 | 0 | 12 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 4 | 0
Neuropathy: sensory (Nervous system disorders) | 1 | 0 | 0 | 4 | 0
Neutrophils/Granulocytes (ANC/AGC) (Investigations) | 1 | 3 | 0 | 14 | 0
Pain (General disorders) | 1 | 1 | 0 | 4 | 0
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 | 1 | 0 | 11 | 0
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0
Prolonged QTc interval (Investigations) | 2 | 0 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 0
AST, SGOT (Investigations) | 0 | 1 | 0 | 8 | 0
Alkaline Phosphatase (Investigations) | 0 | 1 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Cholesterol, high (hypercholestremia) (Investigations) | 0 | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3 | 0
Fever (General disorders) | 0 | 0 | 0 | 3 | 0
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 0 | 3 | 0 | 8 | 0
Lymphocytes (Investigations) | 0 | 2 | 0 | 11 | 0
Nail Changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
PTT (Investigations) | 0 | 1 | 0 | 2 | 0
Pain - Back (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Pain - Joint (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Platelets (Investigations) | 0 | 2 | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0
Amylase (Investigations) | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Glucose, low (hypoglycemia) (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Lipase (Investigations) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT00820170/Prot_SAP_000.pdf